CLINICAL TRIAL: NCT05245890
Title: Assocaiton Between Uric Acid Trajecteries and Remission of Non-alcoholic Fatty Liver Disease (NAFLD) in NAFLD Individuals
Brief Title: Assocaiton Between Uric Acid Trajecteries and Remission of NAFLD in NAFLD Individuals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: The First Afliated Hospital, College of Medicine, Zhejiang University, Hangzhou, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: uric acid trajecteries2022
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Hyperuricemia
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hyperuricemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Uric acid is the end product of dietary or endogenous purines degradation, and hyperuricemia is one of the most common metabolic disorders. A growing body of evidence, comprising a great deal of cross-sectional studies and several prospective ones, also indicates that hyperuricemia is associated with increased prevalence, incidence, and disease severity of non-alcoholic fatty liver disease (NAFLD).

Capitalizing on a cohort study in China, the investigators are aimed to assess the associations of SUA trajecteries with remission of NAFLD in NAFLD individuals and examined whether the association differs across subpopulations.

DETAILED DESCRIPTION:
A cohort study was conducted to evaluate the relationship between the SUA trajecteries and remission of NAFLD. The study enrolled employees who were attending their annual health examination. Furrhermore, the investigators are aimed to explore whether the association differs across subpopulations.

ELIGIBILITY:
Inclusion Criteria:

1. age >=18 years;
2. agree to be enrolled in this study.

Exclusion Criteria:

1. those taking antihypertensive or antidiabetic agents, lipid-lowing agents, or hypouricemic agents;
2. those with alcohol consumption greater than 140 g/week for men and 70 g/week for women;
3. those with a history of other known causes of chronic liver disease such as viral hepatitis or autoimmune hepatitis, and those using hepatotoxic medications.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who undergo annual physical examinations in The First Affiliated Hospital, College of Medicine, Zhejiang University are enrolled in this study. People are divided into two groups according to hepatic ultrasonic examination at baseline: (1) individuals with NAFLD; (2) individuals without NAFLD.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
the severity fatty liver evaluated by hepatic ultrasonic examination | 2 years
  Hepatic ultrasonic examination was performed in all subjects by a trained ultrasonographist who was unaware of the clinical and laboratory data. Hepatic steatosis was diagnosed by characteristic echo patterns according to conventional criteria, such as the evidence of diffuse hyperechogenicity of the liver relative to the kidneys, ultrasound beam attenuation, and poor visualization of intrahepatic structures.

IPD SHARING:
Plan to Share IPD: No